CLINICAL TRIAL: NCT05882630
Title: Surufatinib Combined With Serplulimab Plus Carboplatin and Etoposide as First-line Treatment for Extensive-stage Small-cell Lung Cancer：a Multicenter, Open-label, Phase I/II Trial
Brief Title: Surufatinib Combined With Serplulimab Plus Chemotherapy in the Treatment of Extensive-stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Hunan Cancer Hospital (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-L110
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surufatinib Combined With Serplulimab and EC Chemotherapy (Experimental)
  Interventions: Drug: Surufatinib,Serplulimab,Etoposide,Carboplatin

INTERVENTIONS:
Drug: Surufatinib,Serplulimab,Etoposide,Carboplatin — In dose escalation, Surufatinib will be administered orally (PO) once daily (QD) ,d1-21,q3w + Serplulimab 4.5 mg/kg ivgtt,d1,q3w+Etoposide 100mg/m2,d1-3,q3w + Carboplatin AUC=5,d1,q3w; 4-6 cycles in total.
  At the indication-specific expansion portion of the study, patients will receive surufatinib RP2D,d1-21,q3w+Serplulimab 4.5 mg/kg ivgtt,d1,q3w+Etoposide 100mg/m2,d1-3,q3w + Carboplatin AUC=5,d1,q3w, 4-6 cycles in total. After the end of the first-line treatment, patients with CR, PR, and SD can continue to maintenance treatment with Surufatinib RP2D,d1-21,q3w＋Serplulimab 4.5 mg/kg ivgtt,d1,q3w until the disease progressed.

SUMMARY:
To evaluates the effectiveness and safety of Surufatinib combined with Serplulimab plus chemotherapy for the first-line treatment of ES-SCLC, and maintenance therapy are Surufatinib combined with Serplulimab

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and voluntarily sign informed consent;
2. Age: 18-75 years old;
3. Expected survival period ≥ 3 months;
4. Histologically or cytologically diagnosed with ES-SCLC (Combined small cell lung carcinoma excepted);
5. No prior systemic therapy for ES-SCLC;
6. According to the RECIST 1.1 standard, the patient has at least one target lesion with a measurable diameter;
7. ECOG PS: 0-1;
8. Major organs are functioning well;
9. The urine or serum pregnancy test results of premenopausal women were negative.

Exclusion Criteria:

1. Patients with symptomatic brain metastases;
2. People with hypertension who cannot be well controlled by double antihypertensive drug (systolic blood pressure≥140 mmHg, diastolic blood pressure≥90 mmHg);
3. Urine routine test showed urine protein ≥++ and confirmed 24-hour urine protein quantification>1.0g;
4. Cardiovascular disease history: congestive heart failure> New York Heart Association (NYHA) standard II, patients with active coronary artery disease (those with myocardial infarction 6 months before enrollment can be enrolled), arrhythmia requiring treatment;
5. Active severe clinical infections (>NCI-CTCAE 5.0 version 2 infection criteria), including tuberculosis (clinical evaluation, including clinical history, physical examination, imaging findings and TB examination in line with local clinical practice), hepatitis B (known HBV Surface antigen [HbsAg] positive), hepatitis C or human immunodeficiency virus (HIV 1/2 antibody positive);Patients who have previously had HBV infection or have been cured (defined as the presence of hepatitis B core IgG antibodies and the absence of HBsAg) are eligible. Hepatitis C virus (HCV) antibody-positive patients are only eligible if the HCV RNA polymerase chain reaction is negative.
6. Patients with bleeding tendency or coagulation disorders;
7. In the past 2 years, there are active autoimmune diseases that require systemic treatment (such as corticosteroids or immunosuppressive drugs), and related alternative treatments (such as thyroxine, insulin, or physiological corticosteroid replacement for renal or pituitary insufficiency) are allowed treatment);
8. Patients who are pregnant or breastfeeding;
9. Allergy to any of the drugs in the study;
10. Imaging (CT or MRI) shows that the tumor invades or is poorly demarcated from large vessels;
11. Researchers think it is inappropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival(PFS) | up to 24 months

SECONDARY OUTCOMES:
Objective response rate(ORR) | up to 24 months
Overall Survival(OS) | up to 24 months
Disease control rate(DCR) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No